CLINICAL TRIAL: NCT04730284
Title: Evaluation of a Synbiotic Formula in Patient With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COVSyn
Record Dates: First submitted 2020-08-25; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Coronavirus
Keywords: microbiota
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health supplements (Experimental): One arm only
  Interventions: Other: Health supplements

INTERVENTIONS:
Other: Health supplements — tailor-made Synbiotics, 4g per day for 28 days

SUMMARY:
A series of microbiota were correlated inversely with the disease severity and virus load. Gut microbiota could play a role in modulating host immune response and potentially influence disease severity and outcomes.

DETAILED DESCRIPTION:
Coronavirus can target multiple organs due to the hyperactive immune response with cytokine storms. Several studies have detected SARS-CoV-2 in stool samples and indicated that the virus could spread via faeces. Importantly, COVID-19 uses the same receptor as SARS and this doorway can also be found in the intestine. The cell entry receptor, known as angiotensin converting enzyme 2 (ACE2) receptor mediate entry of SARS-CoV-2 and is highly expressed in small bowel enterocytes. ACE2 is important in controlling intestinal inflammation and its disruption may lead to diarrhoea. In our previous study, stool samples from 15 patients with COVID-19 were analysed. Depleted symbionts and gut dysbiosis were noted even after patients were detected negative of SARS-CoV-2. A series of microbiota were correlated inversely with the disease severity and virus load. Gut microbiota could play a role in modulating host immune response and potentially influence disease severity and outcomes.

In July 2020, there are more than 15 billion confirmed cases globally with 620 thousand deaths. Currently, there are more than 2000 confirmed cases of COVID-19 in Hong Kong. It is important to rebalance the gut microbiota in COVID-19 patients and to improve the symptoms and the quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above; and
2. A confirmed diagnosis of SARS-Cov.2 infection using the PCR according to the standard of according to Centre for Health Protection, Department of Health, HK and released from isolation at recruitment.
3. Written informed consent obtained

Exclusion Criteria:

1. Known allergy or intolerance to the intervention product or its components
2. Any known medical condition that would prevent taking oral probiotics or increase risks associated with probiotics including but not limited to inability to swallow/aspiration risk and no other methods of delivery (e.g., no G/J tube)
3. Known increased infection risk due to immunosuppression such as:

   * Prior organ or hematopoietic stem cell transplant
   * Neutropenia (ANC <500 cells/ul)
   * HIV and CD4 <200 cells/ul
4. Known increased infection risk due to endovascular due to:

   * Rheumatic heart disease
   * Congenital heart defect,
   * Mechanical heart valves
   * Endocarditis
   * Endovascular grafts
   * Permanent endovascular devices such as permanent (not short-term) hemodialysis catheters, pacemakers, or defibrillators
5. Documented pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiome | week 5
  Changes in the gut microbiome (bacteria, virome and fungome) measured by metagenomics at week 5 compared to baseline

SECONDARY OUTCOMES:
Changes in fecal bacteria metabolites | weeks 2, 4, 5, 8 and months 3, 6, 9 and 12
  Changes in fecal bacteria metabolites by PCR at different time points
Change in plasma cytokines including IL-6, IL-IB, TNF-a and CXCL-10 | week 5
  Change in plasma cytokines level at week 5 compared with baseline
Trend in symptom score | weeks 2, 4, 5, 8 and months 3, 6, 9 and 12
  Trend of symptom score at different time points, ranges from 26-104. The higher the score, the worse the symptoms.
Change in Quality of life measured by EQ-5D-5L | weeks 2, 4, 5, 8 and months 3, 6, 9 and 12
  Change in score on Quality of life using EQ-5D-5L at different time points. EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The index can be calculated by deducting the appropriate weights from 1, the value for full health (i.e. state 11111). Each category ranges from 1 to 5. The small the number, the better the health. The EQ-VAS is a vertical visual analogue scale that ranges 0-100 (higher score indicates better imaginable health).
Change in Quality of life measured by SF-12 | weeks 2, 4, 5, 8 and months 3, 6, 9 and 12
  Change in score on Quality of life using SF-12 at different time points. SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. There are formulas for transformation of scale scores so that they will range from 0-100. High score in functioning items indicates better functioning while high score in pain items indicates freedom from pain.
Duration of gastrointestinal symptoms | 4 weeks
  Duration of gastrointestinal symptoms such as anorexia, nausea, vomiting, abdominal pain, bloating within 4 weeks.
Adverse event assessment | 3 months
  Number of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Siew Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Wong CK, Lam CW, Wu AK, Ip WK, Lee NL, Chan IH, Lit LC, Hui DS, Chan MH, Chung SS, Sung JJ. Plasma inflammatory cytokines and chemokines in severe acute respiratory syndrome. Clin Exp Immunol. 2004 Apr;136(1):95-103. doi: 10.1111/j.1365-2249.2004.02415.x. PMID 15030519
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Yeo C, Kaushal S, Yeo D. Enteric involvement of coronaviruses: is faecal-oral transmission of SARS-CoV-2 possible? Lancet Gastroenterol Hepatol. 2020 Apr;5(4):335-337. doi: 10.1016/S2468-1253(20)30048-0. Epub 2020 Feb 20. No abstract available. PMID 32087098
- [Background] Liang W, Feng Z, Rao S, Xiao C, Xue X, Lin Z, Zhang Q, Qi W. Diarrhoea may be underestimated: a missing link in 2019 novel coronavirus. Gut. 2020 Jun;69(6):1141-1143. doi: 10.1136/gutjnl-2020-320832. Epub 2020 Feb 26. No abstract available. PMID 32102928
- [Background] Hashimoto T, Perlot T, Rehman A, Trichereau J, Ishiguro H, Paolino M, Sigl V, Hanada T, Hanada R, Lipinski S, Wild B, Camargo SM, Singer D, Richter A, Kuba K, Fukamizu A, Schreiber S, Clevers H, Verrey F, Rosenstiel P, Penninger JM. ACE2 links amino acid malnutrition to microbial ecology and intestinal inflammation. Nature. 2012 Jul 25;487(7408):477-81. doi: 10.1038/nature11228. PMID 22837003
- [Background] Zuo T, Zhan H, Zhang F, Liu Q, Tso EYK, Lui GCY, Chen N, Li A, Lu W, Chan FKL, Chan PKS, Ng SC. Alterations in Fecal Fungal Microbiome of Patients With COVID-19 During Time of Hospitalization until Discharge. Gastroenterology. 2020 Oct;159(4):1302-1310.e5. doi: 10.1053/j.gastro.2020.06.048. Epub 2020 Jun 26. PMID 32598884
- [Background] WHO Coronavirus Disease (COVID-19) Dashboard. [Assessed on 24 Jul 2020]. https://covid19.who.int/
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Background] Docherty AB, Harrison EM, Green CA, Hardwick HE, Pius R, Norman L, Holden KA, Read JM, Dondelinger F, Carson G, Merson L, Lee J, Plotkin D, Sigfrid L, Halpin S, Jackson C, Gamble C, Horby PW, Nguyen-Van-Tam JS, Ho A, Russell CD, Dunning J, Openshaw PJ, Baillie JK, Semple MG; ISARIC4C investigators. Features of 20 133 UK patients in hospital with covid-19 using the ISARIC WHO Clinical Characterisation Protocol: prospective observational cohort study. BMJ. 2020 May 22;369:m1985. doi: 10.1136/bmj.m1985. PMID 32444460
- [Background] Janowitz T, Gablenz E, Pattinson D, Wang TC, Conigliaro J, Tracey K, Tuveson D. Famotidine use and quantitative symptom tracking for COVID-19 in non-hospitalised patients: a case series. Gut. 2020 Sep;69(9):1592-1597. doi: 10.1136/gutjnl-2020-321852. Epub 2020 Jun 4. PMID 32499303